CLINICAL TRIAL: NCT06650293
Title: Effect of Vitamin D Supplementation as Adjuvant Therapy in Neonatal Jaundice in Combination With Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCHSL-1
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Experimental): Neonates receive phototherapy plus vitamin D
  Interventions: Drug: Vitamin D
- Group-B (No Intervention): Neonates will receive only phototherapy

INTERVENTIONS:
Drug: Vitamin D — Vitamin D supplementation as vitamin D, 2 drops i.e., 800 IU daily for 5 days.
  Arms: Group-A

SUMMARY:
Neonatal jaundice frequently occur during initial week of life. Neonatal jaundice is one of the leading causes of hospital admission and readmission. Some studies have suggested that the healthy newborns with hyperbilirubinemia outside the physiological range have notably reduced serum vitamin D levels. This deficiency is inversely associated with neonatal hyperbilirubinemia, suggesting that low vitamin D levels could be a potential risk factor for jaundice among neonates.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Admitted between 3-28 days of age.
* Indirect hyperbilirubinemia with TSB levels between 14-20 mg/dL
* Born via either cesarean or vaginal delivery
* Birth weight greater than 2500 grams

Exclusion Criteria:

* Prior phototherapy treatment
* Preterm birth (gestational age below 37 weeks).
* SpO2 < 95% at the time of admission
* Severe respiratory distress or failure
* Neonatal sepsis
* Congenital anomalies
* Parents/guardians unwilling to let their neonates be part of this study.

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Total Serum bilirubin levels | 5 days
  Total Serum bilirubin levels evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Zeeshan Afzal, FCPS, Principal Investigator — Pediatric Medicine Department University of Child Health Sciences, Children's Hospital Lahore; Wajiha Rizwan, FCPS, Study Director — Pediatric Medicine Department University of Child Health Sciences, Children's Hospital Lahore
Locations (1):
- Pediatric Medicine Department University of Child Health Sciences, Children's Hospital Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No